CLINICAL TRIAL: NCT02978534
Title: Pharmacokinetics of Quetiapine Across Pregnancy and Postpartum
Acronym: Quetiapine
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Crystal Clark, Assistant Professor, Northwestern University
Other Study IDs: 00201540
Record Dates: First submitted 2016-11-22; First posted 2016-12-01 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Bipolar Disorder
Keywords: pregnant; quetiapine; bipolar; women; female; postpartum; seroquel; perinatal; manic-depressive
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum specimen will be obtained to measure quetiapine and estradiol levels. Standard of care labs will be obtained on every participant that is eligible and signs informed consent. Participants will not have more than 50 ml of blood drawn every 8 weeks. Participants will also have the option to have blood drawn for DNA banking.
  Participants in the study that elect to receive analgesia for pain related to labor and have a spinal-epidural at Northwestern University will have CSF stored and banked for future analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Quetiapine: Patients taking quetiapine during pregnancy are eligible to participate in the study. Their dose and plasma concentration levels of quetiapine will be monitored throughout pregnancy and up to three months postpartum.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — Quetiapine concentrations will be observed in women who have already (under the guidance of a physician) decided to continue taking Quetiapine for the treatment of Bipolar Disorder (any subtype) or Schizophrenia during pregnancy.
  Other Names: Seroquel

SUMMARY:
The widespread and common use of quetiapine in childbearing and pregnant women demands more data to inform dosing and toxicity in pregnancy. The new FDA Pregnancy and Lactation Labeling Final Rule (PLLR) will go into effect on June 30th, 2015 and will replace the prior A, B, C, D, and X categories. Additionally, the PLLR will require information to aid prescribing decisions in three categories 1) Pregnancy (including labor and delivery), 2) Lactation, and 3) Females and Males of Reproductive Potential. The pregnancy category will include a subsection that will describe pharmacokinetic and pharmacodynamic characteristics of the medication in pregnancy, fetal risk, and data quality. The data collected in this study will update the FDA pregnancy pharmacokinetic section for quetiapine and inform physicians that prescribe to childbearing women.

DETAILED DESCRIPTION:
Bipolar Disorder (BD) and Schizophrenia (SCHZ) in pregnancy are associated with pregnancy complications and increased maternal mortality due to physiological and psychosocial changes independent of second-generation antipsychotic (SGA) use. Untreated BD and SCHZ have been associated with an increased risk of placental abnormalities, antepartum hemorrhage, preterm birth, pre-eclampsia, low birth-weight, intrauterine growth retardation, small for gestational age, fetal distress, neonatal hypoglycemia, stillbirth and congenital defects, and the potential for adverse neurodevelopmental outcomes. Severe maternal stress in pregnancy increases the risk for offspring mental disorders, and eye, ear, respiratory, digestive, skin, musculoskeletal, and genitourinary diseases and congenital malformations (i.e., cleft palate, cleft lip). Also, BD and SCHZ illness symptoms are linked to psychosocial consequences that result in poor perinatal outcomes including impulsivity that leads to reckless behavior such as increased indiscriminate sex and exposure to sexually transmitted infections, smoking, increased alcohol and drug use, less prenatal care, and poor nutrition. Furthermore, women with recurrence of mental illness in the perinatal period have increased risk for suicide, a leading cause of maternal death.

The only published case of quetiapine plasma concentrations in a pregnant woman included cross-sectional levels of a woman on 300 mg of quetiapine across pregnancy and postpartum. Compared to six months postpartum, the area under the curve decreased by 27%, 42%, and 18% in the first, second, and third trimester, respectively. Given the complexity of the metabolism of quetiapine to a very active metabolite, it is important to understand the altered metabolism of quetiapine and its active metabolite in pregnancy and the implication for dosing adjustments.

This study will investigate the longitudinal pharmacokinetics of quetiapine in pregnancy, delivery, and postpartum. The long-term goal of this line of research is to establish psychotropic medication dosing algorithms informed by longitudinal pharmacokinetic data to improve mental health and pregnancy outcomes for mothers with serious mental illness.

The primary aims are: 1) Determine the elimination clearance of quetiapine and its major active metabolite, 7-N-desalkyquetiapine, across pregnancy and postpartum; 2) Determine the effect of pharmacokinetic changes on symptoms and toxicity during pregnancy and postpartum, and; 3) Examine the maternal-to-cord plasma concentrations ratios of quetiapine and its major active metabolite, 7-N-desalkylquetiapine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Pregnant, second trimester
* English-speaking
* DSM-V diagnosis of Bipolar Disorder or Schizophrenia, any subtype
* Medically healthy
* Singleton gestation

Exclusion Criteria:

* Chronic use of drugs for medical disorders, except thyroid replacement for stable hypothyroidism
* No psychiatrist or obstetrician
* QIDS-SR 16 positive answer 3 on item 12, "I have made specific plans for suicide or have actually tried to take my life" within the past week
* DSM-V diagnosis of substance abuse or dependence in last 6 months, with the exception of cannabis; positive urine drug screen

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women taking quetiapine for the purpose of mood stabilizing will be recruited broadly from Northwestern clinical services, including Internal Medicine, OB/GYN, Family Medicine, and Psychiatry, registries, and from the local Chicagoland community. Patients that sign consent, complete the evaluation and meet criteria will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-03; Primary Completion 2020-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma concentration/elimination | 2 timepoints during pregnancy (second and third trimesters), and at four and twelve weeks postpartum
  For patients taking the immediate release formulation, plasma levels will be obtained beginning at time 0 and at hours, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 12, 14, 16. For patients on the extended release formulation, plasma levels will be obtained at time 0 and at hours 0.5, 1, 1.5, 2, 2,5, 3, 4, 5, 6, 7, 8, 9, 10, 12, 14, 16, 18, 20, 22, and 24.

SECONDARY OUTCOMES:
Arterial and Venous Umbilical Cord Concentration of Quetiapine and 7-N-desalylquetiapine | 30 minutes
  Arterial and venous cord blood samples will be obtained immediately post-delivery and banked for later analysis
Cerebrospinal Fluid (CSF) Quetiapine and 7-N-desalkyquetiapine Concentrations | CSF to be obtained within 10 minutes of the epidural placement during labor
Scores on Depression assessment, Inventory of Depression Symptomatology- Self Report (IDS-SR) | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum
  To determine if there is a pattern of increasing scores on self-report depression assessment (IDS-SR) and declining plasma levels. Increasing scores indicate worsening symptoms or depression episode recurrence.
Scores on anxiety scale, Generalized Anxiety Disorder (GAD-7) | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum
  To determine if there is a pattern of increasing scores on GAD-7 and declining plasma levels
Scores on mania assessment, Young Mania Reporting Scale (YMRS) | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum.
  To determine if there is a pattern of increasing scores on clinician administered mania assessment (YMRS) and declining plasma levels
Scores on Brief Psychosis Rating Scale (BPRS) | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum.
  assessment to evaluate psychotic symptoms
Positive responses on SAFTEE | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum.
  surveys general and specific side effects including somatic, behavioral, and affective symptoms
Delivery outcomes as determined by the Peripartum Events Scale (PES) | 4 and 12 weeks postpartum
  assessment to quantify stressful events related to delivery.
Scores on the separate domains of the Patient Reported Outcomes Measurement Information System (PROMIS) Global Health | Participants will complete these assessments an average of every 10 weeks from the time they enter the study, up to 12 weeks postpartum.
  Assesses patient perceptions in 5 domains:physical function, pain, emotional distress, social function, and fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal T Clak, MD, MSc, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No